CLINICAL TRIAL: NCT05283252
Title: Evaluating the Effectiveness of Guided Endodontic Microsurgery in Critical Anatomical Structures (A Randomized Clinical Trial)
Brief Title: The 3-Dimensional Printed Guide in Endodontic Microsurgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UDDS-Endo-01-2022
Record Dates: First submitted 2022-02-27; First posted 2022-03-16 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Endodontic Disease; Endodontic Re-treatment Failure
Keywords: Apicoectomy; Guided Endodontic Surgery; Micro-Surgery; Surgical Guide; 3-Dimensional Printed; Critical Structures
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Endodontic Micro-Surgery (Experimental): Use of the 3-D printed guide in endodontic micro-surgery
  Interventions: Device: 3-D printed Guide
- Conventional Endodontic Micro-Surgery (Placebo Comparator): Free-hand endodontic micro-surgery
  Interventions: Other: Conventional Endodontic Micro-Surgery

INTERVENTIONS:
Device: 3-D printed Guide — Guided Endodontic micro-surgery
  Arms: Guided Endodontic Micro-Surgery
Other: Conventional Endodontic Micro-Surgery — Free-hand endodontic micro-surgery
  Arms: Conventional Endodontic Micro-Surgery

SUMMARY:
In recent years, there was a great interest in employing the surgical guide in dentistry due to the development occurred in the 3D printing which became available widely.

Cone beam computed tomography (CBCT) is necessary and crucial in planning for endodontic surgery, but the procedure still depends on how the surgeon reflect the 3D images on the anatomical structures accurately, which may leave room for error.

This study is to compare the clinical and radiographic outcomes using guided endodontic microsurgery versus conventional endodontic microsurgery in critical anatomical structures.

DETAILED DESCRIPTION:
Endodontic microsurgery in critical anatomical structures is considered as a serious challenge for the endodontist.

Major advances have been made to the techniques used in endodontic surgery to make the procedure easier to perform, safer and more predictable.

Several case reports that used surgical guide in endodontic microsurgery found that the procedure was more accurate in control of depth, diameter and angle of osteotomy.

The aim of this study is to compare the clinical and radiographic outcomes using guided endodontic microsurgery versus conventional endodontic microsurgery in critical anatomical structures.

Patients will be selected that they are indicated for endodontic surgery. Upper and lower teeth will be selected close to critical anatomy such as; maxillary sinus, nasal fossa, mental foramen and mandibular canal. medical and dental history will be obtained from all selected patients. Patients will be randomly distributed to either guided micro-surgery group or conventional micro-surgery group. All steps of the surgical procedure will be performed under microscopic magnification. Bioceramic putty will be used as a root-end filling material. Post-surgical instructions will be given to patients. The time of the surgery will be recorded from the first incision to the last suturing. Success and failure will be assessed using radiographic and clinical evaluation at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients in good general health.
* Patients with age ranging between 18-50 years.
* Posterior/anterior teeth close to critical anatomical structures that indicated for endodontic surgery.
* Patients' acceptance to participate in the trail.

Exclusion Criteria:

* Patients with allergy to materials or medications used in the trial.
* Patients with Serious systemic disease incompatible with surgery.
* Pregnant female patients.
* Teeth with periapical pathosis associated with vertical root fracture.
* Non-restorable teeth.
* Teeth with periodontal probe more than 5 mm.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Clinical Success at two weeks | Periodontal tissue healing will be evaluated clinically "2 weeks"
  The position of the oral mucosa at the flap site will be assessed after surgery to evaluate wound healing using the wound healing index (WHI) by Huang et al 2005 as the following criteria:
  Score 1 = uneventful healing with no gingival edema, erythema, suppuration, patient discomfort, or flap dehiscence.
  Score 2 = uneventful healing with slight gingival edema, erythema, patient discomfort, or flap dehiscence, but no suppuration.
  Score 3 = poor wound healing with significant gingival edema, erythema, patient discomfort, flap dehiscence, or any suppuration.
Clinical Success at one year | Clinical signs or symptoms will be evaluated "1 year"
  The patient's symptoms will be evaluated and the examination will be done on percussion, palpation and probing. Clinical Success will be defined as absence of pain, swelling or sensitivity on percussion. Clinical failure is the persistence of any of the above-mentioned symptoms.
Radiographic Success at 6 months | Periapical tissues healing will be evaluated radiographically at 6 months after surgery
  Early follow-up will be done and the initial radiographic Success or failure will be assessed.
  The size of periapical lesions/radiographic transparency will be measured in millimeters by periapical radiographs and CBCT images
Radiographic Success at 12 months | Periapical tissues healing will be evaluated radiographically at 12 months after surgery
  Radiographic Success will be defined as either complete or incomplete healing (formation of scar tissue). Radiographic Failure will involve either uncertain healing (small or constant lesion size) or unsatisfactory healing (increased lesion size).
  The size of periapical lesions/radiographic transparency will be measured in millimeters by periapical radiographs and CBCT images

SECONDARY OUTCOMES:
Time of surgery | During surgery
  The surgical time will be recorded in minutes from the first incision to the last suturing
Change in Pain Perception | Pain will be evaluated at 24, 48, and 72 hours after surgery
  Pain assessment will be performed using a Visual Analog Scale (VAS) which is a subjective measure instrument for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between 0 (no pain) and 10 (worst pain).

CONTACTS AND LOCATIONS:
Overall Officials: Rami Kaddoura, DDS,MSc, Principal Investigator — Damascus University
Locations (1):
- Damascus University, Damascus, Syria

REFERENCES:
- [Background] Buniag AG, Pratt AM, Ray JJ. Targeted Endodontic Microsurgery: A Retrospective Outcomes Assessment of 24 Cases. J Endod. 2021 May;47(5):762-769. doi: 10.1016/j.joen.2021.01.007. Epub 2021 Feb 4. PMID 33548331
- [Background] Lio F, Mampieri G, Mazzetti V, Leggeri A, Arcuri L. Guided endodontic microsurgery in apicoectomy: a review. J Biol Regul Homeost Agents. 2021 May-Jun;35(3 Suppl. 1):47-55. doi: 10.23812/21-3supp1-7. PMID 34289664
- [Background] Popowicz W, Palatynska-Ulatowska A, Kohli MR. Targeted Endodontic Microsurgery: Computed Tomography-based Guided Stent Approach with Platelet-rich Fibrin Graft: A Report of 2 Cases. J Endod. 2019 Dec;45(12):1535-1542. doi: 10.1016/j.joen.2019.08.012. Epub 2019 Oct 9. PMID 31606146
- [Background] Monaghan L, Jadun S, Darcey J. Endodontic microsurgery. Part one: diagnosis, patient selection and prognoses. Br Dent J. 2019 Jun;226(12):940-948. doi: 10.1038/s41415-019-0415-3. PMID 31253911
- [Background] Antal M, Nagy E, Braunitzer G, Frater M, Piffko J. Accuracy and clinical safety of guided root end resection with a trephine: a case series. Head Face Med. 2019 Dec 21;15(1):30. doi: 10.1186/s13005-019-0214-8. PMID 31861995
- [Background] Giacomino CM, Ray JJ, Wealleans JA. Targeted Endodontic Microsurgery: A Novel Approach to Anatomically Challenging Scenarios Using 3-dimensional-printed Guides and Trephine Burs-A Report of 3 Cases. J Endod. 2018 Apr;44(4):671-677. doi: 10.1016/j.joen.2017.12.019. Epub 2018 Feb 14. PMID 29426644
- [Background] Strbac GD, Schnappauf A, Giannis K, Moritz A, Ulm C. Guided Modern Endodontic Surgery: A Novel Approach for Guided Osteotomy and Root Resection. J Endod. 2017 Mar;43(3):496-501. doi: 10.1016/j.joen.2016.11.001. Epub 2017 Jan 28. PMID 28139285